CLINICAL TRIAL: NCT05465603
Title: Rationale for the Use of Elastic Tension Digital Neoprene Orthoses in the Treatment of Proximal Interphalangeal Joint Flexion Contracture: Long Term Results
Brief Title: Rationale and Analysis of the Use of ETDNO in the Treatment of PIPJ Flexion Contracture:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vicenç Punsola Izard (Other)
Responsible Party: Sponsor-Investigator, Vicenç Punsola Izard, Physical Therapist, Certified Hand Therapist in Hand Therapy Barcelona, MSc Gimbernat Universiy , Assistant lecturer at Gimbernat University, PhD Candidate at University of Barcelona, Hand Therapy Barcelona
Organization: Hand Therapy Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Flexion Contracture of Proximal Interphalangeal Joint; Joint Deformities, Acquired
MeSH Terms: conditions — Joint Deformities, Acquired

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients do not know which dose they are reciving compared to the other group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20-22 hours of daily TERT intervention (Experimental): Patients that have suffered an injury to the finger causing flexion contracture of the Proximal interphalangeal joint will be treated using an elastic tension neoprene orthosis for a period of 3 weeks.
  Interventions: Device: ETDNO (Elastic Tension digital neoprene orthosis)
- 11-13 hours daily TERT intervention (Active Comparator): Patients that have suffered an injury to the finger causing flexion contracture of the Proximal interphalangeal joint will be treated using an elastic tension neoprene orthosis for a period of 3 weeks.
  Interventions: Device: ETDNO (Elastic Tension digital neoprene orthosis)

INTERVENTIONS:
Device: ETDNO (Elastic Tension digital neoprene orthosis) — A bespoke orthosis created from neoprene.

SUMMARY:
Introduction: Flexion contracture is one of the most frequent complications in finger trauma. The use of orthoses to obtain the best total end range time (TERT) is the most popular method to treat this pathology . Until now, no orthosis applied for longer than 3 weeks had been able to achieve TERT longer than 12 hours.

Purpose of the study: To assess whether the elastic tension digital neoprene orthosis (ETDNO), using a serial dynamic program, can achieve a better result in ROM and TERT than other orthoses described in the literature.

Methods: analysis of outcomes in a sample of 30 patients with PIP joint flexion contracture treated with the ETDNO and serial dynamic program.

DETAILED DESCRIPTION:
In this study the researcher will compare the efect of daily TERT treatment on the proximal interphalangeal joint contracture using an ETDNO. The investigator will treat two different groups one with a dose of from 11 to 13 hours of the ETDNO while the other one is treated with a dose of from 20 to 22 hours of daily TERT with the same device. This treatment will last three weeks and will be evalauted the first day, the he first week and the third week. At the end of the study the researcher will quantify the improvement on both groups to know which dailyTERT dose is the best option.

ELIGIBILITY:
Inclusion Criteria:

* PIP flexion contracture

Exclusion Criteria:

* more than 6 month of contracture and more than 45º of flexion contracture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Extension improvement | 3 weeks
  The degree of extension of the PIP at the end of the treatment compared with the beginning

CONTACTS AND LOCATIONS:
Overall Officials: Vicenç Punsola-Izard, Principal Investigator — Hand Therapy Barcelona
Locations (1):
- Hand Therapy Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
will be available in the papers published